CLINICAL TRIAL: NCT02641041
Title: A Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB033 in Healthy Japanese Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of BIIB033 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 215HV102; 2015-004560-11 (EudraCT Number)
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Central Nervous System (CNS) Demyelinating Disease; Multiple Sclerosis
Keywords: Japanese; Single Ascending Dose (SAD); Multiple Ascending Dose (MAD)
MeSH Terms: conditions — Demyelinating Diseases; Multiple Sclerosis | interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): A single IV dose of 10 mg/kg BIIB033 or placebo given on Day 1
  Interventions: Biological: BIIB033; Other: Placebo
- Cohort 2 (Experimental): A single IV dose of 30 mg/kg BIIB033 or placebo given on Day 1
  Interventions: Biological: BIIB033; Other: Placebo
- Cohort 3 (Experimental): One IV dose of 100 mg/kg BIIB033 or placebo given on Days 1 and 15
  Interventions: Biological: BIIB033; Other: Placebo

INTERVENTIONS:
Biological: BIIB033 — single or multiple dose
Other: Placebo — single or multiple dose

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of a single dose and multiple doses of BIIB033 administered to healthy adult Japanese participants. The secondary objectives of this study are to evaluate the pharmacokinetics (PK) profile of BIIB033 administered as single and multiple doses in healthy adult Japanese participants and to assess the single-dose and multiple-dose immunogenicity of BIIB033.

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese subjects must have been born in Japan, and their biological parents and grandparents must all have been of Japanese origin.
* Subjects who have lived out of Japan for more than 5 years must not have significantly modified their diets since leaving Japan.
* Must be a nonsmoker or light smoker (<10 cigarettes per day) and be willing to abstain from using tobacco and tobacco-containing products during the Inpatient Period and for at least 48 hours prior to Day -1, Day 14 (for Cohort 3), and all outpatient visits.
* Must have a body mass index of 18 to 32 kg/m2, inclusive.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* Serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within the 3 months prior to Day -1.
* Fever or bacterial or viral infection (including upper respiratory tract infection) within 2 weeks prior to Day -1.
* History of severe allergic or anaphylactic reactions.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to day 113
Number of participants with clinically significant laboratory parameters | Up to day 113
Number of participants with clinically significant vital sign abnormalities | Up to day 113
Number of participants with clinically significant electrocardiograms (ECGs) abnormalities | Up to day 113
Number of participants with clinically significant physical examination abnormalities | Up to day 113
Number of participants with clinically significant neurological examination abnormalities | Up to day 113

SECONDARY OUTCOMES:
PK parameter of BIIB033: Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to day 113
PK parameter of BIIB033: Area under the concentration-time curve from time zero to the time of the last measurable sample (AUClast) | Up to day 113
PK parameter of BIIB033: AUC over a given dosing interval | Up to day 113
PK parameter of BIIB033: Maximum observed concentration (Cmax) | Up to day 113
PK parameter of BIIB033: Time to reach maximum observed concentration (Tmax) | Up to day 113
PK parameter of BIIB033: Terminal elimination half-life (t1/2) | Up to day 113
PK parameter of BIIB033: Volume of distribution at steady state (Vss) | Up to day 113
PK parameter of BIIB033: Clearance (CL) | Up to day 113
PK parameter of BIIB033: accumulation ratio (RAC) | Up to day 113
Number of participants with positive serum BIIB033 antibodies | Up to day 113

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, West Yorkshire, United Kingdom